CLINICAL TRIAL: NCT05050383
Title: Drug-Induced Sleep Endoscopy (DISE): Phenotyping Obstruction Patterns
Brief Title: DISE: Phenotyping Obstruction Patterns
Acronym: DISE-PhOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Raj Dedhia, MD, Associate Professor, Director of Sleep Surgery, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 849542
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea; drug-induced sleep endoscopy; snoring
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Drug-Induced Sleep Endoscopy (Other): Drug-Induced Sleep Endoscopy
  Interventions: Other: Pharyngeal Manometry; Other: Submental Ultrasound

INTERVENTIONS:
Other: Pharyngeal Manometry — Catheters will be passed into the nose and advanced to the pharynx to measure airway pressures during drug-induced sleep.
Other: Submental Ultrasound — Ultrasound of airway soft tissues

SUMMARY:
Drug-induced sleep endoscopy (DISE) represents an opportunity to evaluate the upper airway in sleep-like conditions. In its current clinical form, however, DISE does not routinely determine the functional impact of anatomic and neuromuscular factors on airflow obstruction.

The investigators will apply nasal pressure (CPAP) during DISE to generate pressure-flow and pressure-area relationships, deriving functional determinants of upper airway obstruction during sleep. In addition, they will use objective anatomic measurements from computerized tomography (CT) and submental ultrasound. The findings will allow the investigators to streamline the upper airway exam during DISE, and will further the goal of developing personalized solutions that address specific pathogenic mechanisms of pharyngeal collapse and airflow obstruction during sleep.

The investigators will use the physiologic and anatomic features derived from DISE and imaging to determine which are predictive of success to standard-of-care surgical interventions (e.g. skeletal, soft tissue, neurostimulation) .

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized by recurrent upper airway obstruction due to inadequate muscle tone during sleep leading to nocturnal hypercapnia, repeated oxyhemoglobin desaturations and arousals. Continuous positive airway pressure (CPAP) is the therapeutic mainstay for OSA, but adherence remains poor.

Currently, there exist 3 classes of surgical therapy for OSA, each addressing a specific pathologic structure: skeletal surgery (target: jaw bones), neurostimulation (target: tongue), and soft tissue (target: soft palate). Unfortunately, there is a critical knowledge gap in terms of accurately identifying a patient's underlying mechanism of obstruction; as a result, the efficacy of surgical treatment is limited.

Drug-induced sleep endoscopy (DISE) represents an opportunity to evaluate the upper airway in sleep-like conditions. In its current clinical form, however, DISE does not routinely determine the functional impact of anatomic and neuromuscular factors on airflow obstruction. In June 2020, the investigators implemented a pilot protocol (IRB # 833511) to utilize measures of airflow, pressure catheters, and ultrasound to enhance DISE exams. Over the course of 100 patients, they refined the research protocol to generate a safe, efficient, and comprehensive physiologic exam of the upper airway in the clinical setting (Dedhia et al, ORL, 2021, in press).

Upper airway pressure-flow and pressure-area relationships will be characterized during a standard-of-care DISE by stepping through a range of nasal pressure (CPAP) levels to derive functional determinants of upper airway obstruction during sleep. The investigators' preliminary work in this area has shown patients requiring lower pressures to restore airflow experience improved outcomes with neurostimulation surgery. Their overall hypothesis is that upper airway pressure-flow/area relationships can be used to predict response to all 3 major classes of sleep surgery: skeletal, neurostimulation, and soft tissue. They will address this hypothesis by characterizing upper airway pressure-flow and pressure-area relationships while utilizing objective anatomic measurements from CT and ultrasound. These findings will allow investigators to streamline the upper airway exam during DISE, and will further the goal of developing personalized solutions that address specific pathogenic mechanisms of pharyngeal collapse and airflow obstruction during sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 18yrs) willing and capable of providing informed consent.
2. English-speaking & able to give Informed Consent.
3. Referred or scheduled for clinically indicated DISE procedure.
4. Seeking CPAP alternatives for treatment of sleep disordered breathing.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Identify the pathogenic determinants of airway obstruction at specific sites of pharyngeal collapse by characterizing upper airway pressure-flow/area relationships during DISE to predict responses to upper airway surgery | Within 1 year of enrollment
  Change in pre-operative to post-operative AHI

SECONDARY OUTCOMES:
Correlation of anatomic measurements from computerized tomography (CT) scans to physiologic findings from DISE | Within 3 months of enrollment
  Craniofacial measurements of bones and soft tissues from CT scans
Complement videoendoscopic DISE findings with synchronous ultrasound imaging | Within 3 months of enrollment
  Ultrasonic evaluation of dynamic tongue motion during DISE
Compare positive airway pressure levels obtained from natural sleep to those during DISE | Within 3 months of enrollment
  Therapeutic CPAP levels
Examine outcomes associated with non-surgical treatments (e.g. oral appliance therapy) | Within 1 year of enrollment
  Polysomnography metrics (e.g., apnea:hypopnea ratio), questionnaire data (ESS, ISI, FOSQ-10, NOSE, Snoring VAS, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Raj C Dedhia, MD, MSCR, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No